CLINICAL TRIAL: NCT06364813
Title: Co-developing a Novel Intervention to Promote Wellbeing of Family Caregivers of Individuals With Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Somayyeh Mohammadi, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H20-01461
Record Dates: First submitted 2024-02-15; First posted 2024-04-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries; Caregiver Burden
Keywords: Caregiving; eHealth; online education; family caregivers
MeSH Terms: conditions — Spinal Cord Injuries; Caregiver Burden

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMPANION Group (Experimental): eHealth education: participants receive family caregiving education through the COMPANION eHealth program.
  Interventions: Other: COMPANION eHealth Program
- No Intervention (No Intervention): Control group participants will receive the usual care available at their local rehabilitation clinic.

INTERVENTIONS:
Other: COMPANION eHealth Program — COMPANION consists of online, self-paced educational modules with information on a range of topics such as providing medical care, applying for financial aid and home aid, working on the relationship with the care recipient, dealing with mental health issues, and learning life skills.
  Arms: COMPANION Group

SUMMARY:
Family caregivers of individuals with spinal cord injury (SCI) provide the majority of care and are at high risk of experiencing caregiver burden, which not only impacts caregivers' own wellbeing, but also their ability to respond to patients' needs. Health education using online approaches (eHealth) has the potential to improve quality of care, enhance communication between health care users and providers, reduce costs and increase access to existing knowledge and education for family caregivers. Here, the investigators propose a research study to assess the quality of the eHealth program. The findings of this study will lead to the refinement of the eHealth program.

DETAILED DESCRIPTION:
People with spinal cord injury (SCI) experience an irreversible neurological impairment. Each year there are more than 17,000 and 3,500 new cases of SCI in the United States and Canada, respectively. The estimated lifetime health care and direct economic cost that SCI imposes is between $1.6m and $3m (CAD) per person. However, this number is substantially higher when unpaid care provided by family caregivers is considered. Family caregivers of individuals with SCI provide the majority of care, from assistance with activities of daily living to managing finances. Family caregivers report negative social and health-related consequences such as difficulties in maintaining a social life or full-time employment. Family caregivers also tend to ignore their own mental and physical health needs. The burden and distress caused by caregiving responsibilities not only impacts caregivers, but also caregivers' ability to respond to the patients' needs. Therefore, it is essential to better understand and address the needs and challenges faced by family caregivers. In preliminary work conducted to explore these issues, the investigators examined the needs and challenges of family caregivers of individuals with SCI through conducting a systematic review, an online survey and semi-structured interviews. Working with end-users partners and building on this line of research, the investigators aim to provide the information and resources required and requested by family caregivers to address their needs via an eHealth tool. Through this needs-based technology intervention, the investigators' goal is to improve the physical and psychological wellbeing of family caregivers of individuals with SCI and, ultimately, to improve the well-being of the individuals with SCI. In addition, the investigators will investigate patterns of health care use among family caregivers and individuals with SCI as a means to evaluate the impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Family caregiver of an adult individual with SCI
* Must be older than 18 years old
* Must live in Canada
* Must live with the individual with SCI in the community
* The spinal cord injury of the individual with SCI must have happened no earlier than 6 months prior to participation

Exclusion Criteria:

* Family caregiver with major medical and physical conditions that needs routine visits to medical doctors (e.g., cancer)
* Family caregivers of individuals with SCI who are still in a rehabilitation facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Family caregivers' subjective burden as assessed by the Zarit Burden Interview | 0 months, 3 months, and 6 months
  The 12-item Zarit Burden Interview uses a 5-point scale to measure family caregivers' subjective burden by asking participants how often they experience certain feelings. Individual responses range from 0 (never) to 4 (nearly always) and are added to generate a total score. Total scores can range from a minimum of 0 to a maximum of 48. A total score ranging between 0-10 indicates no to mild burden, 10-20 indicates mild to moderate burden, and >20 indicates high burden. The Zarit Burden Interview will be administered via survey at 3 timepoints.

SECONDARY OUTCOMES:
Participants' objective burden as assessed by the Dutch Objective Burden Inventory | 0 months, 3 months, and 6 months
  The 38-item Dutch Objective Burden Inventory will be used to measure family caregivers' objective burden by assessing participants' perceived burden relating to care activities over the past three months. Individual responses are scored (1 = Not at all burdensome, 2 = somewhat burdensome, 3 = very burdensome) and the average calculated to produce a total score (ranging from 1 to 3). Higher averages indicate higher objective burden. The Dutch Objective Burden Inventory will be administered via survey at 3 timepoints.
Participants' distress as assessed by the Depression, Anxiety and Stress Scale | 0 months, 3 months, and 6 months
  The Depression, Anxiety and Stress Scale (DASS) contains 21 items assessing distress over the past week using a 4-point Likert scale (0=never, 3=always). Responses for each item will be scored and averaged into a single distress indicator with higher scores indicating more distress. The DASS will be administered via survey at 3 timepoints.
Participants' relationship quality satisfaction as assessed by the Dyadic Adjustment Scale | 0 months, 3 months, and 6 months
  The Dyadic Adjustment Scale (DAS-32) consists of 32 items for measuring the level of relationship quality satisfaction among dyads in general and during the past few weeks. Total scores range from 0 to 151. Higher scores indicate less distress and high adjustment. The DAS-32 will be administered via survey at 3 timepoints.
Participants' health-related quality of life as assessed by the Veterans RAND 12-item Health Survey | 0 months, 3 months, and 6 months
  The Veterans RAND 12-item Health Survey (VR-12) is a questionnaire that will be used to measure family caregivers' health-related quality of life during the past four weeks and compared to their health one year ago. Items relate to general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health. 2 separate scores are generated from responses, a "Physical Health Summary Measure (PCS-physical component score)" and a "Mental Health Summary Measure (MCS-mental component score)". The VR-12 scoring algorithm is used to score PCS and MCS based on weights derived from 877,775 responses to a Veterans RAND 36-Item Health Survey (VR-36) that was administered federally to American veterans in 1999, resulting in variable minimum and maximum score values. Higher PCS and MCS scores indicate better health. The VR-12 will be administered via survey at 3 timepoints.
Caregiver competence as assessed by the Caregiving Competence Scale | 0 months, 3 months, and 6 months
  Caregiver competence is measured by a 4-item Likert scale asking participants to rate feelings about their competency and performance of their caregiving role. Response options range from 4 = "very much" to1 = "not at all". Total score values range from 0 to 12 with higher scores indicating higher caregiving competence. The Caregiving Competence Scale will be administered via survey at 3 timepoints.
Caregiver costs as assessed by the Caregiver Indirect and Informal Care Cost Assessment Questionnaire | 0 months, 3 months and 6 months
  The Caregiver Indirect and Informal Care Cost Assessment Questionnaire (CIIQ) consists of 13 items with information including, but not limited to, work status, time missed at work, productivity, and physical and emotional caregiving duties. Responses are open-ended apart from one item using a 10-point scale ranging from 0 ("could work as usual") to 10 ("Could not work at all"). Calculations will be conducted to estimate indirect and informal caregiver costs. Total scores report cost in dollars and can range from as low as zero to any maximum number. Higher scores indicate greater financial impact due to informal care costs. The CIIQ will be coupled with a bespoke item asking about additional money fcSCI spend on themselves. To minimize concerns about recall, a one-week recall period will be used for the CIIQ and a three-month recall period will be used for the bespoke item.
Participants' opinion regarding the usability of the implementation as assessed by the System Usability Scale | 3 months and 6 months
  The System Usability Scale (SUS) consists of a 10-item questionnaire with five response options scored on a Likert scale ranging from "Strongly agree" to "Strongly disagree." It is used to measure usability of the eHealth implementation based on participants' experience using COMPANION over the last 3 months. It will be administered only to participants in the intervention group via survey at 2 timepoints. Raw scores range from 0-40 and are algorithmically converted into meaningful SUS scores ranging from 0-100. Higher scores indicate higher perceived usability.
Participants' experience using the implementation as assessed by a qualitative interview | 6 months
  Optional semi-structured interviews (45-60 minutes) will be used to explore fcSCI's experience with the eHealth implementation. Interview guides will be created to ask participants to share their perspective on advantages and disadvantages of the program. Participating in the interview will only be offered to participants in the intervention group.

OTHER OUTCOMES:
A composite measure of recruitment rate, consent rate, retention rate, perceived benefit, and assessor masking will be evaluated as "successful" or "revise" according to expectations | Through study completion, an average of 6 months
  Recruitment rate will be successful if a total of 40 participants and a mean of 3-4 participants per month are recruited. Consent rate will be successful if <10% of participants refuse to consent. Retention rate will be considered successful if >80% of participants complete data collection at 6 months. Perceived benefit will be assessed by responses to the System Usability Scale (at 3 months and 6 months) and the qualitative interview at 6 months, and will be successful if >85% of responses to the SUS are "strongly agree/agree", and if analysis of interview responses will inform clinical importance. Assessor masking will be considered successful if 100% of participants do not unmask their treatment to the study assessor. The evaluation of these feasibility indicators will be used to assess process issues in the study protocol.
A composite measure of treatment adherence, participant and evaluator burden during data collection, and expert burden will be evaluated as "successful" or "revise" according to expectations | Through study completion, an average of 6 months
  Treatment adherence will be considered successful if >85% of participants complete all the modules in COMPANION. Participant and evaluator burden will be considered successful if (i) >85% of participants complete baseline data collection (at 0 months) in ≤2 hours, and (ii) >85% of participants complete data collection at 3 months and 6 months in ≤1.5 hours. Expert burden will be considered successful if (i) the mean time spent per participant is <2 hours during the first 3 months of the study, (ii) the mean time spent per participant is <1 hour during the following 3 months of the study, and (iii) research staff make follow-up phone calls for clarification with <20% of participants. The evaluation of these feasibility indicators will be used to assess resource issues in the study protocol.
A composite measure of internet stability, participant processing time, and treatment administration issues will be evaluated as "successful" or "revise" according to expectations | Through study completion, an average of 6 months
  Internet stability will be assessed by reported downtime from accessing COMPANION due to technical or mechanical issues and will be considered successful if more than 90% of participants are not without internet for more than 2 days. Participant processing time will be assessed by time passing from data collection to treatment and will be considered successful if the mean time between data collection and accessing treatment is less than 10 days at initial data collection (0 months) and data collection at 3 months. Treatment administration issues will be assessed by study educator responses to a post-treatment evaluation form and will be considered successful if any issues identified through the evaluation form are deemed modifiable without requiring substantial changes to the study protocol. The evaluation of these feasibility indicators will be used to assess management issues in the study protocol.
A measure of dose level of training time | Through study completion, an average of 6 months
  Dose level (e.g., time spent in the education modules) response will be assessed by the correlation between time spent (in minutes) using the module and change in burden scores. It will be considered successful if there is a positive correlation. The evaluation of these feasibility indicators will be used to assess treatment issues in the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, PhD, Study Chair — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammadi S, Erlander B, Cathcart H, Robillard JM, Sauvageau S, Whitehurst DGT, Pauly E, Page B, Miller WC. Codeveloping a Novel Intervention to Promote the Well-Being of Family Caregivers of Individuals With Spinal Cord Injury: Protocol for a Feasibility Randomized Control Trial. JMIR Res Protoc. 2025 Sep 25;14:e67709. doi: 10.2196/67709. PMID 40998319